CLINICAL TRIAL: NCT05861856
Title: Comparison of the Efficiency of Manual Therapy and Virtual Reality Supported Core Stabilization Exercises in Patient With Adolescent Idiopathic Scoliosis
Brief Title: Manual Therapy and Virtual Reality Supported in Patient With Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Eylem KÜÇÜK, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HacettepeUEK
Record Dates: First submitted 2023-05-07; First posted 2023-05-17 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent idiopathic scoliosis; Manual therapy; Virtual reality; Core stabilization exercises
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality group (Active Comparator): Virtual reality supported core stabilization exercises will be performed.
  Interventions: Other: Virtual reality
- Manual therapy group (Active Comparator): Mobilization for the spine, mobilization and relaxation methods for the soft tissues around the spine will be performed.
  Interventions: Other: Manual therapy
- Combine group (Active Comparator): Both virtual reality supported core stabilization exercises and manual therapy techniques will be applied.
  Interventions: Other: Manual therapy; Other: Virtual reality

INTERVENTIONS:
Other: Manual therapy — Mobilization for the spine, mobilization and relaxation methods for the soft tissues around the spine will be performed.
  Arms: Combine group; Manual therapy group
Other: Virtual reality — Virtual reality supported core stabilization exercises will be performed.
  Arms: Combine group; Virtual reality group

SUMMARY:
Adolescent Idiopathic Scoliosis is a three-dimensional deformity of the trunk and spine of unknown cause seen in adolescents. There are various conservative treatment methods to treat scoliosis. Manual therapy and exercises are a few of these treatments. There are studies showing that manual therapy reduces the severity of curvature, increases range of motion, modulates tissue/muscle extensibility, improves soft tissue movement limitation, relieves pain, and increases psychological well-being in scoliosis patients. In order to treat scoliosis, there are various exercise applications that are applied specifically to scoliosis, from physiotherapy applications. Core stabilization is one of the exercise methods that aim to keep the spine in the center.

Virtual reality, on the other hand, is a three-dimensional simulation model that gives its participants the feeling of reality and allows mutual communication with a dynamic environment created by computers. Virtual reality is a method that provides the opportunity to work with task-based techniques by creating stimulating and entertaining environments, using people's interests and motivations. In a study, it was stated that two of the scoliosis-specific exercises were done through video-assisted games, but they stated that there was no difference because the number of exercises was low. Therefore, in this study, it was aimed to apply core stabilization exercises to scoliosis patients with virtual reality application and to investigate their effects on recovery in patients. In addition, it is planned to investigate whether the severity of the curvature in patients decreases further and whether it has an effect on other healing parameters by using the virtual reality treatment application together with manual treatment.

DETAILED DESCRIPTION:
Male and female volunteer patients who were diagnosed with "Adolescent Idiopathic Scoliosis" and referred to physical therapy and met the inclusion criteria will be included in the study. Patients whose families and themselves agreed to participate voluntarily in this study will be randomly divided into three groups and included in the study. Virtual reality supported core stabilization exercises (stability enhancing exercises for the muscles around the spine), manual therapy (mobilization for the spine, mobilization and relaxation methods for the soft tissues around the spine) techniques for the second group, and both virtual reality supported core stabilization exercises and exercises for the third group were given to the third group. Manual therapy techniques will also be applied. The treatment program was planned as a total of 16 sessions, 2 days a week for 8 weeks. This study was planned as single-blind for the purpose of impartiality of the evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AIS
* Age 10-16 years
* Cobb angle was between 10° and 25
* Risser sing did not exceed 4
* Informed consent forms were signed by the parents and children

Exclusion Criteria:

* Used brace,
* Had previous spinal surgery, inferior limb length difference,
* Could not exercise due to another injury/diagnosis,
* Had neuromuscular, psychiatric, cardiovascular, respiratory insufficiency and mental disability

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2023-07-29 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-11-12 (Actual)

PRIMARY OUTCOMES:
Cobb angle | Change from pretreatment and 8 weeks after treatment.
  The most accepted way of scoliosis evaluation is Cobb angle measurement performed on frontal plane x-ray. The Cobb angle is the curvature of the spine, and measuring it is essential for determining the severity of scoliosis, selecting the best course of action, and monitoring the progression or regression of cases following treatment. The Cobb angle measure as the vertically intersecting angle after determining the vertebrae above the apex and below the apex, which are the most tilted from the concave side of the curvature of the spine.
Angle of Trunk Rotation | Change from pretreatment and 8 weeks after treatment.
  It assessed with a Bunnell scoliometer is a type of inclinometer that measures the asymmetry of the degree of axial rotation on both sides of the body. Assessment is in a standing, forward-bending position bent-over position (arms dangling, palms pressed together) with the pelvis horizontal, and subject standing on a foot template

SECONDARY OUTCOMES:
Walter Reed Visual Assessment Scale | Change from pretreatment and 8 weeks after treatment.
  It was designed to measure physical deformity as perceived by patients with idiopathic scoliosis. The scale assesses seven aspects of the deformity: spinal curvature, rib prominence, flank prominence, deformity/alignment of the thorax with respect to the pelvis, trunk imbalance, shoulder asymmetry and scapular asymmetry. Scores for each catagory range from 1 (no deformity) to 5 (the worst deformity), and the total score is generated from the sum of the scores from the seven domains.
Scoliosis Research Society-22 | Change from pretreatment and 8 weeks after treatment.
  Scale is a simple and practical quality of life questionnaire specially created for individuals with scoliosis. SRS includes parameters such as pain, self-image/appearance, function/activity, mental health, and satisfaction with treatment. It is also stated that it is effective in evaluating the changes that occur with treatment. The questionnaire has a total of 22 items that are scored from 1 (worst) to 5 (best) for each item.

CONTACTS AND LOCATIONS:
Overall Officials: Eylem Küçük, Principal Investigator — Amasya University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years
Access Criteria: upon request